CLINICAL TRIAL: NCT00880711
Title: Faslodex International Observational Non-Interventional Study in Advanced Breast Cancer
Brief Title: Faslodex International Observational Non-Interventional Study in Advanced Breast Cancer (BC)
Acronym: FIONA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OAT-FAS-2009/1
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: Fiona; Faslodex; Advanced Breast Cancer; Real life data; Collect real life data in clinical practice across Austria
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patient with advanced BC, already receiving Faslodex therapy

SUMMARY:
The purpose is to collect real life data on the use of fulvestrant in normal clinical practice in Austria and document the clinical benefit of fulvestrant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with hormone receptor-positive locally advanced or metastatic breast cancer
* Ability to read and write and complete questionnaires
* Provision of written informed consent
* Patients who already received a prescription for fulvestrant

Exclusion Criteria:

* A subject who does not fulfil all the above mentioned inclusion criteria is not allowed to participate in this NIS

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitals, office based specialists
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit, defined as the development of at least one of the following stages and holding on for at least 6 month: Complete response, partial response or stable disease | Baseline, after 3, 6, 9 month

SECONDARY OUTCOMES:
Tolerability | After 3, 6, 9 month (as per usual clinical practice)
Quality of Life | Baseline, after 3, 6, 9 month (as per usual clinical practice)
Performance status (Karnofsky Index) | Baseline, after 3, 6, 9 month (as per usual clinical practice)

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Steger, Univ Prof. Dr., Study Chair — Medical University of Vienna
Locations (13):
- Austria (13):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Leoben
  - Research Site, Linz
  - Research Site, Oberpullendorf
  - Research Site, Rankweil
  - Research Site, Rottenmann
  - Research Site, Salzburg
  - Research Site, Sankt Veit im Pongau
  - Research Site, Steyr
  - Research Site, Vienna
  - Research Site, Wiener Neustadt